CLINICAL TRIAL: NCT01599026
Title: Cardiac Septal Hypertrophy in the Fetus of Diabetic Mother and Its Effect on Postnatal Cardiac Function
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, heba mohamed, Cardiac septal hypertrophy in the fetus of diabetic mother and its effect on postnatal cardiac function, Ain Shams Maternity Hospital
Other Study IDs: dhvf 7531
Record Dates: First submitted 2012-05-14; First posted 2012-05-15 (Estimated); Last update posted 2012-05-15 (Estimated); Status verified 2012-05

CONDITIONS: Cardiology in Fetus of Diabetic Mother
Keywords: cardiology; fetus of diabetic mother

STUDY DESIGN:
Time Perspective: Cross-Sectional

SUMMARY:
Good glycemic control is superior to poor glycemic control in reducing risk of interventricular septum thickness among fetuses of diabetic mothers

DETAILED DESCRIPTION:
Good glycemic control is superior to poor glycemic control in reducing risk of interventricular septum thickness among fetuses of diabetic mothers specially during third trimester of pregnancy

ELIGIBILITY:
Inclusion Criteria:

* singleton pregnancy
* gestational age 36 weeks

Exclusion Criteria:

* congenital anomalies
* obstetric complications
* medical disorders other than diabetes

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: diabetic pregnant ladies gestational age more than 35 weeks
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2012-04; Primary Completion 2013-02 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
To study interventricular septum thickness in fetus of diabetic mother and correlate it with good glycemic control. | one year
  To study interventricular septum thickness in fetus of diabetic mother and correlate it with good glycemic control during third trimester of pregnancy.

SECONDARY OUTCOMES:
cardiac function in infant of diabetic mother | one year
  To correlate postnatal cardiac function to interventricular septum thickness to reach cut of value of septum thickness for prenatal prediction of symptomatic cardiomyopathy in infant of diabetic mother.

CONTACTS AND LOCATIONS:
Locations (1):
- AinShamsMH, Cairo, Egypt